CLINICAL TRIAL: NCT01316367
Title: Effectiveness of PRECEDE Model for Health Education on Cardiovascular Risk Reduction in Patients With Type 2 Diabetes Mellitus
Brief Title: Effectiveness of PRECEDE Model for Health Education on Changes and Level of Control in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Carlos III, Madrid (Other)
Responsible Party: Miguel Ángel Salinero Fort, Hospital Carlos III
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCIII-0106; PI02-0567 (Other Grant/Funding Number: Fondo de Investigación Sanitaria)
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2003-03

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Risk Factor
Keywords: Health Promotion Education; Type 2 Diabetes Mellitus; Cardiovascular Risk Factors; Spain
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Health Promotion Education (CHPE). (Active Comparator): The CHPE model was defined according to the recommendations of the Spanish Ministry of Health National Conference on Diabetes Mellitus, which was complemented by criteria for good care of the Madrid Primary Healthcare Service for the promotion of healthy lifestyles among adults (2004-2007). The model is based on the following aspects: self-monitoring of glycaemic control, physical exercise, diet, weight management, and times of the day when the patient was most vulnerable to overeating, and given improved understanding of the relative effects of certain food choices on blood glucose control, medication adherence and smoking cessation.
  Interventions: Behavioral: CHPE
- PRECEDE HPE model (Experimental)
  Interventions: Behavioral: PRECEDE HPE model

INTERVENTIONS:
Behavioral: PRECEDE HPE model — The model considers the influence of the following three factors on health-related behavior:
  * Predisposing: factors influencing the patient's motivation to undertake the behavior to be analyzed or encouraged.
  * Facilitators: factors influencing the level of easiness or difficulty the patient and his/her family have in undertaking a given behavior.
  * Reinforcing: factors arising after the patient has undertaken the behavior, and which reward or punish it.
  Arms: PRECEDE HPE model
Behavioral: CHPE — The CHPE model was defined according to the recommendations of the Spanish Ministry of Health National Conference on Diabetes Mellitus, which was complemented by criteria for good care of the Madrid Primary Healthcare Service for the promotion of healthy lifestyles among adults (2004-2007). The model is based on the following aspects: self-monitoring of glycaemic control, physical exercise, diet, weight management, and times of the day when the patient was most vulnerable to overeating, and given improved understanding of the relative effects of certain food choices on blood glucose control, medication adherence and smoking cessation.
  Arms: Conventional Health Promotion Education (CHPE).

SUMMARY:
BACKGROUND: Individual health education is considered to be essential in the overall care of patients with type 2 diabetes (DM2), although there is some uncertainty regarding its metabolic control benefits. There have been very few randomized studies on the effects of individual education on normal care in DM2 patients with a control group, and none of these have assessed the long-term results. Therefore, this study aims to use this design to assess the effectiveness of the PRECEDE (Predisposing, Reinforcing, Enabling, Causes in Educational Diagnosis, and Evaluation) education model in the metabolic control and the reduction of cardiovascular risk factors, in patients with type 2 diabetes.

METHODS: An open community randomized clinical trial will be carried out in 8 urban community health centers in the Northeastern Madrid (Spain). Six hundred patients with DM2 will be randomized in two groups: PRECEDE or conventional model for health promotion education. The main outcome measures is glycated hemoglobin A1C, body mass index (BMI), blood pressure, lipids and control criteria during the 2-year follow-up period.

DETAILED DESCRIPTION:
Assignment to the Health Promotion Education (HPE) will be random, three centers will use conventional HPE (the control group) and the remaining five will use PRECEDE-type HPE. Eligible patients are selected from a list of DM2 patients by each professional using random sampling, until the predetermined sample size is attained.

Conventional HPE is defined according to the recommendations of the Spanish Ministry of Health National Conference on Diabetes Mellitus, and was complemented by the criteria for good care of the Madrid Primary Healthcare Service for the promotion of healthy lifestyles among adults for 2004-2007

ELIGIBILITY:
Inclusion Criteria:

* Older than 30 years of age, with previously diagnosed DM2 (cardinal clinical, plus random blood glucose > 200 mg/dl or oral glucose of > 200 mg/dl at 2 h, twice, or plasma fasting glucose of > 126 mg/dl on two occasions or being diagnosed previously, received specific treatment for DM2)

Exclusion Criteria:

* Gestational diabetes
* Patients involved in clinical trials
* Patients with life expectancy less than 1 year (according to clinical judgment)
* Patients who refused to participate
* Homebound patients Patients meeting criteria for inclusion and not meeting any exclusion criteria were invited to participate, and were included after accepting and signing an informed consent form.

Min Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2003-02; Primary Completion 2005-02 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
HbA1c level | Final (before 2 years follow-up)

SECONDARY OUTCOMES:
Blood Pressure | Final (before 2 years follow-up)
  Systolic and Diastolic Blood Pressure
Low-density lipoprotein (LDL) cholesterol | Final (before 2 years of follow-up)
Body Mass Index (BMI) | Final (before 2 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Salinero, MD, Principal Investigator — Hospital Carlos III, Madrid
Locations (1):
- Hospital Carlos III, Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Salinero-Fort MA, Carrillo-de Santa Pau E, Arrieta-Blanco FJ, Abanades-Herranz JC, Martin-Madrazo C, Rodes-Soldevila B, de Burgos-Lunar C. Effectiveness of PRECEDE model for health education on changes and level of control of HbA1c, blood pressure, lipids, and body mass index in patients with type 2 diabetes mellitus. BMC Public Health. 2011 Apr 28;11:267. doi: 10.1186/1471-2458-11-267. PMID 21524316